CLINICAL TRIAL: NCT07180394
Title: Botulinum Toxin for Strabismus Treatment
Acronym: Botox Squint
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Ayesha Saeed, Public Health Officer, Foundation University Islamabad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUMCRCT2; 1004/RC/FFH/RWP (Other Grant/Funding Number: Fauji Foundation Hospital, Rwp)
Record Dates: First submitted 2025-08-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Strabismic Deviation; Strabismus
Keywords: Strabismus; esotropia; exotropia; hypotropia; hypertropia; Botulinum toxin; therapy; outcomes
MeSH Terms: conditions — Strabismus; Esotropia; Exotropia

STUDY DESIGN:
Intervention Model Description: The primary objective is to examine the efficacy and outcomes of Botox (botulinum toxin) intramuscular injection therapy in the treatment of pediatric or adult strabismus
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botulinum toxin for strabismus treatment (Experimental): The primary objective is to examine the efficacy and outcomes of Botox (botulinum toxin) intramuscular injection therapy in the treatment of pediatric or adult strabismus
  Interventions: Drug: Botox injection into extraocular muscles

INTERVENTIONS:
Drug: Botox injection into extraocular muscles — Botulinum toxin in various doses by injecting it into the overacting extraocular musces in strabismus patients, especially pediatric, but also adult cases, to use it as an alternative for strabismus surgery. For children, it will be administered under sedation or general anesthesia and in adults, under topical anesthesia. The pre-operative measurements of the type of strabismus, patterns, deviation, and post-operative results will be studied both in the short and long-term.

SUMMARY:
The bacterial species Clostridium botulinum produces a class of neurotoxins known as botulinum toxin. At the neuromuscular junction, botulinum toxin A prevents acetylcholine from being released. Following a Botox intramuscular injection, the injected EOM becomes paralysed 2-4 days after the injection and remains so clinically for at least 5-8 weeks. Muscle function recovery takes five to fourteen weeks, depending on the injection site, volume, and concentration of the solution, as well as the innervation density.

Botulinum toxin treatment results in a pharmacologic recession of the injected extraocular muscle, and the muscle lengthens while its agonist contracts, paralysing it. Improved ocular alignment or a decrease in the severity of the deviation may last for a long time, even if the pharmaceutical impact normally goes away after three months.

Even after the pharmacologic effect has worn off, a number of elements, such as mechanical, proprioceptive, and binocular effects, may intervene during the period of muscle paralysis to help stabilise and improve alignment in strabismus patients over the long term.

DETAILED DESCRIPTION:
Detailed Description: A Strabismus or squint is an ocular condition characterized by misalignment of the eyes. It derived from the Greek word "strabismos" meaning 'to look obliquely'. It can be categorized as congenital or acquired, based on onset; by direction; as concomitant or incomitant/paralytic; and as isolated or syndromic. The prevalence of strabismus in the general population ranges from 2-5%, with a lower prevalence of 0.6% observed in the Asian population.

Normal ocular alignment depends upon the integrity of the extraocular muscles, orbital connective tissues, cranial nerves supplying these muscles, fusion centers, and the visual cortex. The etiopathogenesis of strabismus involves abnormalities in binocular vision or neuromuscular control of ocular motility. Left untreated and unrecognized, strabismus can result in irreversible visual impairment, amblyopia, and abnormalities with binocular vision. Moreover, it can significantly impact the affected individual's personality and lead to undesirable cosmetic concerns, such as misdirected eyes, abnormal facial and head posture, and occasionally, peculiar eye movements like up-shoots or down-shoots. It also has psychosocial implications for those affected by it.

The standard therapy for strabismus is either correction of the refractive errors causing it or strabismus surgery under general anesthesia in our country. For optimal benefit, adjustable strabismus surgery is done for cooperative children and adults. This requires 4-6 hours for the general anesthesia to be worn off and may not be an option for very small children and babies, for whom optimal results may not be obtained, in addition to long general anesthesia time.

For more than thirty years, botulinum toxin A has been utilised as a pharmaceutical treatment for strabismus. The majority of the literature on strabismus views it primarily as a surgical substitute, contingent on the strabismologist's preference. But as time and experience have shown, Botulinum toxin is not just an alternate treatment; it also has some other indications in which surgery is not a smart choice. Although there are few randomised controlled trials, Botulinum toxin appears to work similarly to surgery for certain motility issues. Botulinum toxin produces a "chemodenervation" effect, inhibits the release of acetylcholine, and tampers with calcium metabolism. The paralytic effect lasts for two months after injection into an EOM, with the maximal effect occurring in five to seven days. BTXA's overall weakening impact lasts for six to nine months. It is anticipated that the antagonist will experience a relative contraction when under the influence of Botulinum toxin.

Although Botulinum toxin has a short-term impact on extraocular muscles (EOM), it may lead to a long-term reduction in deviation. Potential explanations for this long-lasting effect could include changes in the number of sarcomeres during its effect, immunohistochemical modifications, and central adaptive mechanisms that show up as better binocularity.

The primary goal of this study is to examine the efficacy and outcomes of botulinum toxin intramuscular injection therapy in the treatment of pediatric or adult strabismus, instead of performing surgery in these patients.

Our plan to use the Botulinum toxin in various doses by injecting it into the overacting extraocular musces in strabismus patients, especially pediatric, but also adult cases, to use it as an alternative for strabismus surgery. For children, it will be administered under sedation or general anesthesia and in adults, under topical anesthesia under sterile aseptic techniques. The preoperative and postoperative measurements of the type of strabismus, patterns, deviation, and post-operative results will be studied both in the short and long-term.

ELIGIBILITY:
Inclusion Criteria:

* Esotropia or exotropia presenting with a small-to-moderate angle deviation (<40 PD)

  * Acute onset comitant esotropia
  * Postoperative residual or consecutive strabismus (2-8 weeks postoperatively or later)
  * Acute paralytic strabismus to alleviate diplopia while the palsy resolves (mainly sixth nerve palsies, sometimes fourth nerve palsy)
  * Active thyroid eye disease (Graves Disease), inflamed or pre-phthisical eyes, when surgery is not recommended
  * Adjunct to surgery for large-angle esotropia or sixth nerve palsy or for large-angle exotropia
  * As a muscle sparing option in patients at risk of anterior segment ischemia

Exclusion Criteria:

* Unrealistic expectations

  * Neuromuscular disorders: Amyotrophic Lateral Sclerosis (ALS), Myasthenia Gravis and Eaton-Lambert syndrome
  * Pregnancy and breastfeeding

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Strabismus Angle in Prism Diopters (PD) in the Primary Position from the baseline angle at Week 2, Week 6, 3 months, 6 months, 9 months, and 1 year of the first intramuscular botox injection. | Baseline, at 2 weeks post injection, to 1 year post injection
  Using the prism cover test (PCT), the strabismus angle in the primary position was determined. The mean of the strabismus angle when viewed from a distance of 6 meters and when viewed from a distance of 33 centimetres was used to calculate the strabismus angle. The same afflicted eye (either the left or the right) was used for each participant's examination for the course of the trial. The difference between the values at Week 2, Week 6, 3 months, 6 months, 9 months, and 1 year and baseline, was used to compute the change from Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sana Nadeem Assoc. Prof., FCPS, Principal Investigator — Foundation University Islamabad
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
the data may be made available in the public repository, or on request from PI

REFERENCES:
- [Background] Badakere A, Badrinath V, Dhillon HK, Valliappan A, Natarajan V, Agarkar S. Botulinum toxin A as a treatment modality for acute acquired comitant esotropia - An Indian perspective. Indian J Ophthalmol. 2025 Feb 1;73(2):228-230. doi: 10.4103/IJO.IJO_2198_23. Epub 2024 Aug 14. PMID 39186638
- [Background] Scott AB, Fahn S, Brin MF. Treatment of strabismus and blepharospasm with Botox (onabotulinumtoxinA): Development, insights, and impact. Medicine (Baltimore). 2023 Jul 1;102(S1):e32374. doi: 10.1097/MD.0000000000032374. PMID 37499080
- [Background] Bort-Marti AR, Rowe FJ, Ruiz Sifre L, Ng SM, Bort-Marti S, Ruiz Garcia V. Botulinum toxin for the treatment of strabismus. Cochrane Database Syst Rev. 2023 Mar 14;3(3):CD006499. doi: 10.1002/14651858.CD006499.pub5. PMID 36916692